CLINICAL TRIAL: NCT06843200
Title: Conversations With Caregivers About Health and Appearance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00001483
Record Dates: First submitted 2025-01-30; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-01

CONDITIONS: Disordered Eating Behaviors; Depression; Feeding Behaviors; Parent-Child Relations
MeSH Terms: conditions — Disordered Eating Behavior; Depression; Feeding Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): a single 2-hour, remote delivered interactive group parenting session
  Interventions: Behavioral: Parent Group Discussion
- Wait-list control (No Intervention): wait-list control group will receive the same intervention after data collection ends

INTERVENTIONS:
Behavioral: Parent Group Discussion — A 2-hour interactive parent group delivered to 5-10 parents via zoom; discuss weight bias and discrimination; brainstorm ways to respond in parent-child interactions involving health and appearance; and identify action steps.
  Arms: Intervention

SUMMARY:
This clinical trial is evaluating the effects of a 2-hour, small group discussion with parents and caregivers of adolescents in Oregon. We will evaluate whether parents'/caregivers' experience reductions in their disordered eating symptoms, mood symptoms, and parent-child relationship quality, relative to parent/caregiver participants in the wait list control. We will also evaluate whether the children of these parents/caregivers experience improvements in their disordered eating and mood symptoms.

ELIGIBILITY:
Inclusion criteria for parent/caregiver:

* at least 18 years old
* the primary caregiver of at least one child 12-17 years old who lives with them at least 50% of the time
* living in the state of Oregon
* can read and understand English at the 6th grade level or higher
* access to internet and private space for zoom

Inclusion criteria for the child:

* 12-17 years of age
* can read and understand English at the 6th grade level or higher

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Parent/caregiver disordered eating symptoms | baseline to 1-month
  Disordered eating will be measured using the 36-item Eating Disorder Examination Questionnaire (EDE-Q)
Parent-child feeding practices | baseline to 1-month
  Child feeding practices will be assessed using the modified Comprehensive Feeding Practices Questionnaire (CFPQ). The monitoring, restriction for weight, restriction for health, environment, modeling, and teaching about nutrition subscales (27-items) will be used. 4 responses on the measure are rated on a 5-point scale from 1 (never) to 5 (always), while the rest are rated on a 5-point scale from 1 (disagree) to 5 (agree).
Parent/caregiver weight bias internalization | baseline to 1-month
  Weight bias internalization will be measured using the modified 10-item Weight Bias Internalization Scale (WBIS-M). Responses on the measure are rated on a 7-point scale from 1 (strongly disagree) to 7 (strongly agree).
Exercise avoidance | baseline to 1-month
  Exercise avoidance will be assessed using 2-items used in previous research (More et al., 2019). Responses on the measure are rated on a 7-point scale from 1 (not at all true) to 7 (completely true).
Parent/caregiver self-compassion | baseline and 1-month
  Self-compassion will be assessed using the 12-item Self-Compassion Scale-Short Form (SCS-SF). Responses on the measure are rated on a 5-point scale from 1 (almost never) to 5 (almost always). Higher summed scores indicate greater self-compassion. The SCS-SF has near perfect correlation with the original 26-item Self-Compassion Scale.
Parent/child body ideal internalization | baseline and 1-month
  Sociocultural attitudes towards appearance, including thin-ideal internalization, muscular-ideal internalization, and appearance-related pressures will be measured using three subscales from the Sociocultural Attitudes Towards Appearance Questionnaire Revised-3 (SATAQ-R). The Internalization-TV/Mag, Internalization-Athlete, and Internalization-Comparison subscales (13-items) subscales will be used. Responses on the measures are rated on a 5-point scale from 1 (definitely disagree) to 5 (definitely agree).
Parent/caregiver stress | baseline and 1-month
  Parental stress will be measured using the 18-item Parental Stress Scale (PSS). Responses on the measure are rated on a 5-point scale from 1 (strongly disagree) to 5 (strongly agree).
Parent/caregiver fat talk | baseline and 1-month
  Frequency of fat talk will be assessed using the 16-item Family Fat Talk Questionnaire. Responses on the measure are rated on a 5-point scale from 1 (never) to 5 (always).
Parent/caregiver anti-fat attitudes | baseline and 1-month
  Anti-Fat attitude will be assessed using 3-items from the Willpower subscale of the Anti-Fat Attitudes Questionnaire (AFA). Responses on the measure are rated on a 9-point scale from 0 (very strongly disagree) to 9 (very strongly agree).

SECONDARY OUTCOMES:
child disordered eating symptoms | baseline to 1-month
  Disordered eating will be measured using the 36-item Eating Disorder Examination Questionnaire (EDE-Q).
Parent-child relationship (child report) | baseline to 1-month
  Child perceived quality of relationship with parent will be measured using the 8-item Parent-Adolescent Relationship Scale. Three items on the measure are rated on a 5-point scale from 0 (strongly disagree) to 4 (strongly agree) while the other 5 items on the measure are rated on a 5-pooint scale from 0 (never) to 4 (always). This measure has been validated in an adolescent sample.
child anti-fat bias | baseline to 1-month
  Anti-Fat attitude will be assessed using 3-items from the Willpower subscale of the Anti-Fat Attitudes Questionnaire (AFA). Responses on the measure are rated on a 9-point scale from 0 (very strongly disagree) to 9 (very strongly agree). This measure has been validated in an adolescent sample.
Child exercise avoidance | baseline to 1-month
  Exercise avoidance will be assessed using 2-items used in previous research (More et al,, 2019). Responses on the measure are rated on a 7-point scale from 1 (not at all true) to 7 (completely true).
fat talk (child report of parent/caregiver) | baseline and 1-month
  Frequency of fat talk will be measured using the 14-item Fat Talk Questionnaire. Responses on the measure are rated on a 5-point scale from 1 (never) to 5 (always). Our team will make revisions to the language in the scale to replace gendered language with gender neutral language. This measure has been validated in adolescents 12 and up.
child weight bias internalization | baseline and 1-month
  Weight bias internalization will be measured using the modified 10-item Weight Bias Internalization Scale (WBIS-M). Responses on the measure are rated on a 7-point scale from 1 (strongly disagree) to 7 (strongly agree). The measure has been validated in an adolescent sample.
child body ideals internalizations | baseline and 1-month
  Sociocultural attitudes towards appearance, including thin-ideal internalization, muscular-ideal internalization, and appearance-related pressures will be measured using three subscales from the Sociocultural Attitudes Towards Appearance Questionnaire Revised-3 (SATAQ-R). The Internalization-TV/Mag, Internalization-Athlete, and Internalization-Comparison subscales (13-items) subscales will be used. Responses on the measures are rated on a 5-point scale from 1 (definitely disagree) to 5 (definitely agree). This measure has been validated in an adolescent sample.
child self-compassion | baseline and 1-month
  Self-compassion will be assessed using the 17-item Self-Compassion Scale Youth Version (SCS-Youth). Responses on the measure are rated on a 5-point scale from 1 (almost never) to 5 (almost always). Higher summed scores indicate greater self-compassion. The SCS-Youth has been validated in an adolescent sample.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oregon, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No